CLINICAL TRIAL: NCT03081767
Title: Comparison of Standard PET/CT vs. Digital PET/CT
Brief Title: Standard PET/CT vs. Digital PET/CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Andrei Iagaru, Chief of the Division of Nuclear Medicine and Molecular Imaging, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB Protocol: 39329
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-03

CONDITIONS: Cancer
Keywords: PET/CT; digital PET/CT
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Patients undergoing digital PET/CT (Other): Single arm prospective study of paired imaging studies. Patients who are referred to Nuclear Medicine and are scheduled to undergo imaging on the standard PET/CT will also have imaging performed on the digital PET/CT.
  Interventions: Diagnostic Test: Digital PET/CT scan

INTERVENTIONS:
Diagnostic Test: Digital PET/CT scan — The Division of Nuclear Medicine and Molecular Imaging at Stanford has installed the first ever GE-made digital PET/CT scanner worldwide. The investigators wish to determine if the digital PET/CT scanner offers equivalent image quality as the standard PET/CT scanner.

SUMMARY:
The investigators wish to determine if standard and digital PET/CT scanners provide equivalent results for disease detection and diagnosis.

DETAILED DESCRIPTION:
There will be a single injection of the PET radiopharmaceutical followed by a standard PET/CT scan and immediately after by the digital PET/CT scan, or vice versa. The investigators wish to determine if image quality is equivalent with the digital PET/CT scanner.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years old at the time of the scan
* Patient provides written informed consent
* Patient is referred for standard (F18 FDG; F18 NaF; Ga68 DOTATATE) or research (68Ga PSMA or 68Ga RM2) PET/CT
* Patient is capable of complying with study procedures
* Patient is able to remain still for duration of imaging procedure (approximately 60 minutes total for both PET/CT)

Exclusion Criteria:

* Patient is pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Iagaru, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duan H, Baratto L, Hatami N, Liang T, Mari Aparici C, Davidzon GA, Iagaru A. 68Ga-PSMA11 PET/CT for biochemically recurrent prostate cancer: Influence of dual-time and PMT- vs SiPM-based detectors. Transl Oncol. 2022 Jan;15(1):101293. doi: 10.1016/j.tranon.2021.101293. Epub 2021 Nov 22. PMID 34823095
- [Result] Baratto L, Toriihara A, Hatami N, Aparici CM, Davidzon G, Levin CS, Iagaru A. Results of a Prospective Trial to Compare 68Ga-DOTA-TATE with SiPM-Based PET/CT vs. Conventional PET/CT in Patients with Neuroendocrine Tumors. Diagnostics (Basel). 2021 May 30;11(6):992. doi: 10.3390/diagnostics11060992. PMID 34070751

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Undergoing Digital PET/CT: Patients referred to Nuclear Medicine undergo imaging on the standard positron emission tomography/computed tomography (PET/CT) and also have imaging performed on the digital PET/CT.
Period: Overall Study
Arm/Group | Patients Undergoing Digital PET/CT
Started | 199
Completed | 199
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients Undergoing Digital PET/CT: Patients referred to Nuclear Medicine undergo imaging on the standard PET/CT and also have imaging performed on the digital PET/CT.
Arm/Group | Patients Undergoing Digital PET/CT
Number analyzed (Participants) | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 144
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 176
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 1
  White | 159
  More than one race | 0
  Unknown or Not Reported | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 199

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Image Quality
Description: Diagnostic image quality will be determined using a 5-point Likert Scale that reads:
  5 - Diagnostic: Excellent diagnostic image quality;
  4 - Diagnostic: Good diagnostic image quality;
  3 - Diagnostic: Acceptable diagnostic image quality;
  2 - Sub-optimal diagnostic: image quality with limited additional clinical information;
  1 - Non-diagnostic: non-diagnostic image quality
Time Frame: an expected average of 3 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Digital PET/CT: Imaging using digital PET/CT.
- Standard PET/CT: Imaging using standard PET/CT.
Arm/Group | Digital PET/CT | Standard PET/CT
Number analyzed (Participants) | 199 | 199
score on a scale | 4.96 (0.20) | 4.30 (0.47)
Statistical Analysis 1: Comparison: Digital PET/CT vs Standard PET/CT; Test type: Other; p < 0.0000001, t-test, 2 sided — Actual P-Value = 3.89597E-42. A P-value of <0.05 was considered significant

ADVERSE EVENTS:
Time Frame: 1 day (average approximately 3 hours).
Arm/Group | Digital PET/CT | Standard PET/CT
All-Cause Mortality (participants affected / at risk) | 0/199 | 0/199
Serious Adverse Events (participants affected / at risk) | 0/199 | 0/199
Other Adverse Events (participants affected / at risk) | 0/199 | 0/199

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT03081767/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT03081767/SAP_001.pdf